CLINICAL TRIAL: NCT05658861
Title: Comparing the Gastric Transit of Commercial Milk Containing A1 Beta-casein and A2 Milk Containing Only A2 Beta-casein Using Magnetic Resonance Imaging (MRI)
Brief Title: Comparing the Gastric Transit of Commercial Milk and A2 Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Dennis A. Savaiano, Professor, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: IRB-2019-296
Record Dates: First submitted 2022-12-07; First posted 2022-12-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Lactose Intolerance, Adult Type
MeSH Terms: conditions — Lactose Intolerance, Adult Type

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Milk containing A1 and A2 beta-casein — Single dose of commercial milk
  Other Names: Commercial milk
Other: Milk containing only A2 beta-casein — Single dose of A2 milk
  Other Names: A2 milk

SUMMARY:
Cow's milk contains two types of β-casein: A1 and A2. The μ-opioid peptide BCM-7 is released from A1 but not from A2. BCM-7 is associated with slower gastrointestinal transit and hence increased gastrointestinal transit times. Lactose maldigesters reported an increase in abdominal pain due to consumption of milk containing A1 beta-casein as compared to milk containing only A2 beta-casein. The hypothesis of this study is that the differential abdominal pain is due to the differential gastric transit. This is a double-blinded, randomized, controlled trial conducted to determine if the transit of A1 β-casein milk is modified in the stomach as compared to milk with only A2 β-casein.

DETAILED DESCRIPTION:
Recruitment:

Flyers, emails, and advertisements in local and university newspapers will be used for recruitment of study participants.

Phone screening:

Interested individuals will be contacted via phone by study staff to assess eligibility by asking questions listed in the inclusion and exclusion criteria.

Informed consent:

If the individual is eligible through phone screening, the study staff will read and explain the informed consent to the individual. Informed consent will contain all the information regarding study procedure, compensation, risks and benefits. If Informed Consent is granted, the participant will be contacted through their preferred method of contact (email or phone) to schedule a hydrogen breath test (HBT).

Screening lactose maldigesters via HBT:

Maldigestion will be classified by a rise of breath hydrogen concentration of greater than 20ppm after a challenge dose of 2% commercial milk containing 0.5g lactose per kg body weight. Participants will consume a low-fiber meal and then fast 12 hours prior to HBT. A breath sample will be obtained from participants just before drinking the milk dose. Participants will then consume milk containing 0.5 grams lactose per kilogram body weight. Breath samples will be obtained according to the following schedule: 0 hour (pre dose), 30 minutes, 1 hour, 90 minutes, 2 hours, 3 hours, 4 hours, 5 hours and 6 hours. Participants who exhibit a rise of breath hydrogen concentration of greater than 20ppm between any two timepoints of the 6-hour test will be classified as lactose maldigesters, and will be qualified to enter the intervention portion of the study.

Intervention:

There will be two in-person visits in intervention.

Visit 1:

Participants should fast for 12 hours and avoid consuming water for 3 hours prior to the MRI scanning appointment. On the day of the visit, participants will undergo a safety screening for MRI compatibility as required by the Purdue MRI Facility and Inner Vision West. Prior to MRI scanning, all participants will remove any metal objects and change into medical scrubs provided by the facility. Participants will then consume their first randomized milk containing 0.5 grams lactose per kilogram body weight (Upper limit - 0.5g/kg up to 50g of lactose). Images of the stomach will be obtained at 0 (pre dose/baseline), 10, 30, 60 and 120 minutes using a Magnetom 3T Prisma MRI scanner. Participants will rate their abdominal pain at 0, 30, 60, 90 and 120 minutes.

Visit 2:

There will be at least a 6-day interval between Visit 1 and Visit 2. The same procedure from visit 1 will be followed in visit 2. Participants will consume the second randomized milk containing 0.5 grams lactose per kilogram body weight during this visit.

ELIGIBILITY:
Inclusion Criteria:

* Ability/desire to provide informed consent
* Aged 18 to 65 years of age inclusive at screening
* Milk intolerant and identified as a lactose maldigester while participating in the Milk Protein Study (applicable only for subjects from the previous milk protein study and not applicable for new subjects)
* Current or recent history of intolerance to or avoidance of dairy of at least one month duration (by self-report and self-reported symptoms).
* Willing to return for all study visits and complete all study related procedures
* Able to understand and provide written informed consent in English

Exclusion Criteria:

* • Currently pregnant

  * Diagnosed with any of the following disorders known to be associated with abnormal gastrointestinal motility such as; Gastroparesis, amyloidosis, neuromuscular diseases (including Parkinson's disease), collagen vascular diseases, alcoholism, uremia, malnutrition, or untreated hypothyroidism
  * History of surgery that alters the normal function of the gastrointestinal tract including, but not limited to: gastrointestinal bypass surgery, bariatric surgery, gastric banding, vagotomy, fundoplication, pyloroplasty [Note: history of uncomplicated abdominal surgeries such as removal of an appendix more than 12 months prior to screening will not be excluded]
  * Past or present : Organ transplant, chronic pancreatitis, pancreatic insufficiency, symptomatic biliary disease, Celiac disease, chronic constipation, diverticulosis, inflammatory bowel disease (IBD), ulcerative colitis (UC), Crohn's disease (CD), small intestine bacterial overgrowth syndrome (SIBO), gastroparesis, gastro-esophageal reflux disease (GERD), Irritable Bowel Syndrome (IBS) or any other medical condition with symptoms that could confound collection of adverse events.
  * Active ulcers, or history of severe ulcers
  * Diabetes mellitus (type 1 and type 2)
  * Congestive Heart Failure (CHF)
  * Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C
  * Recent use of systemic antibiotics defined as use within 30 days prior to screening
  * Any of the following: Worked with metal (grinding, fabrication, etc.) or had an injury to the eye involving a metallic object (e.g., metallic slivers, foreign body, been injured by a metallic object that may NOT have been completely removed (e.g., bullets, shrapnel, BBs), had a reaction to a contrast medium used for MRI or CT, have claustrophobia (fear of closed places), been diagnosed with epilepsy/seizure, any reason you would be unable to remain still for long periods of time, Cardiac pacemaker, Any type of prosthesis (eye, penile), Implanted cardiac defibrillator, Heart valve prosthesis/stents, Aneurysm clip, Shunt (spinal/intraventricular), Neuro or Bone Stimulator, Wire sutures or surgical staples, Insulin or Infusion Pump, Bone/joint pin, screw, nail, plate, Implanted drug infusion device, Body tattoos, Cochlear, otologic or ear implant, Tattooed makeup (eyeliner, lip, etc.), Prostate radiation seeds, Breast tissue expander, IUD (intrauterine device), Hearing aids, Transdermal medicine patch (Nitro),Body piercing(s), Any metallic implants or objects, any other reason the participant thinks they would not be a good candidate for MRI.
  * Any other conditions/issues noted by the study staff and/or Principal Investigator that would impact participation and/or protocol compliance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Volume of milk in stomach/gastric transit | 2 hours
  Volume of milk in the stomach will be calculated using FSL software with MRI images acquired at 0, 10, 30, 60 and 120 minutes.

SECONDARY OUTCOMES:
Difference in abdominal pain | 2 hours
  Abdominal pain will be rated using a 6-point Likert Scale. The scale ranges from a score of 0 to 5 (0 = none, 1 =slight, 2 = mild, 3 = moderate, 4 = moderately severe, 5 = severe).

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Savaiano, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue MRI Facility, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jianqin S, Leiming X, Lu X, Yelland GW, Ni J, Clarke AJ. Effects of milk containing only A2 beta casein versus milk containing both A1 and A2 beta casein proteins on gastrointestinal physiology, symptoms of discomfort, and cognitive behavior of people with self-reported intolerance to traditional cows' milk. Nutr J. 2016 Apr 2;15:35. doi: 10.1186/s12937-016-0147-z. PMID 27039383
- [Background] Ramakrishnan M, Eaton TK, Sermet OM, Savaiano DA. Milk Containing A2 beta-Casein ONLY, as a Single Meal, Causes Fewer Symptoms of Lactose Intolerance than Milk Containing A1 and A2 beta-Caseins in Subjects with Lactose Maldigestion and Intolerance: A Randomized, Double-Blind, Crossover Trial. Nutrients. 2020 Dec 17;12(12):3855. doi: 10.3390/nu12123855. PMID 33348621